CLINICAL TRIAL: NCT07039721
Title: Intestinal Hyperechogenicity Confirmed by Evaluation of Gray Spectra
Acronym: HICE Spectre
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL25_0422
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-06

CONDITIONS: Echogenicity; Intestinal Foetus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Evaluation of echogenicity: Patients ongoing a routine 2nd or 3rd trimester ultrasound will have an extra 5 minutes of ultrasound with a specifc intestinal setting
  Interventions: Other: Evaluation of echogenicity

INTERVENTIONS:
Other: Evaluation of echogenicity — Patients ongoing a routine 2nd or 3rd trimester ultrasound will have an extra 5 minutes of ultrasound with a specific intestinal setting

SUMMARY:
Hyperechoic bowel is an ultrasound anomaly observed in screening and diagnostic ultrasound, and associated with various fetal pathologies including cystic fibrosis, chromosomal abnormalities, maternal-fetal infections (notably Cytomegalovirus CMV) and intrauterine growth retardation. Suspicion of hyperechogenic intestines in a fetus during a screening ultrasound leads to referral of the mother to a specialized antenatal diagnostic consultation. If the diagnosis is confirmed, this may lead to further investigations, including genetic analyses, which are costly for the healthcare system. However, many of the patients referred after a screening examination for this reason actually have their diagnosis invalidated during the specialized consultation. These "false alarms" lead to an overload of specialist consultations, and are a source of concern for couples.

. However, many of the patients referred after a screening examination for this reason actually have their diagnosis invalidated during the specialist consultation. These "false alarms" lead to an overload of specialist consultations, and are a source of concern for couples.

The diagnosis of intestinal hyperechogenicity is difficult because it is based on the sonographer's subjective impression, with a 3-grade gradation according to the echogenicity of the intestine in relation to the bone (Slotnick and Abuhamad. 1996). According to this method, the evaluation is carried out by progressively decreasing the gain applied to the image: if the hyperechoic bowel disappears before the iliac bone, it's a grade 1; if the bowel and iliac bone disappear at the same time, it's a grade 2; and finally if the bowel is still visible on the image while the iliac bone has disappeared, it's a grade 3.

In addition to gain, which, if too high, tends to overestimate the diagnosis of hyperechoic bowel, other ultrasound parameters can vary the subjective impression of bowel echogenicity, such as the use of high-frequency probes or the application of harmonics, which also lead to overdiagnosis (Lee and Cho. 2003).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* in the second and third trimesters of pregnancy,
* singletons or twins, diamniotics, adults,
* undergoing screening or diagnostic ultrasound at obstetric and gynecology department,
* on the Samsung Hera W10 ultrasound machine during the study
* Patient able to understand the ins and outs of the study
* Patient has been informed of the study and has expressed no objection to participating in it.

Exclusion Criteria:

* Minor patients
* Persons deprived of their liberty by judicial or administrative decision
* Persons under psychiatric care
* Persons admitted to a health or social institution for purposes other than research
* Adults under legal protection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — study carried out on pregnant patients
Study Population: This study focuses on patient followed for their routine exam during their 2nd or 3rd trimester of pregnancy at the Gynecology and obstetric ward of the Femme-Mere-Enfant Hospital of the Hospices Civils de Lyon
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Grey level comparison | At inclusion
  The gray levels measured on the fetal intestines will be compared before and after the application of a pre-established "intestines" adjustment program to the same patient carrying a healthy fetus during an ultrasound scan performed in the second or third trimester of pregnancy, by producing two gray level histograms covering two groups of pixels contained in 10x10mm ellipses containing either the fetal intestines or part of the fetal bone.
  The histograms obtained are associated with a greyscale average, provided by the camera. We will calculate the ratio between the average grey levels of the intestines and the bone, before and after applying the settings.
  The aim is therefore to compare, quantitatively and accurately, the gray levels at intestinal and bone levels in second- and third-trimester fetuses, before and after the application of specific presettings.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Edouard Herriot, Lyon, Rhone, France